CLINICAL TRIAL: NCT01907594
Title: Effects of Nicotine Replacement Therapy and D-cycloserine on Nicotine Treatment Seekers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Ran out of funding
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, S. Rob Vorel, Principal Investigator, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 6769
Record Dates: First submitted 2013-07-10; First posted 2013-07-25 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Cycloserine; Nicotine Replacement Therapy; Transdermal Patch; Autogenic Training

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- D-cycloserine (Active Comparator): The investigators will randomize participants to either DCS 250 mg or placebo, administered daily for four days.
  Interventions: Drug: D-cycloserine; Drug: Nicotine Replacement Therapy (patch); Behavioral: Smoking Cue Exposure; Behavioral: Progressive Muscle Relaxation
- Gelatin Capsule (Placebo Comparator): The investigators will randomize participants to either DCS 250 mg or placebo, administered daily for four days.
  Interventions: Drug: Nicotine Replacement Therapy (patch); Behavioral: Smoking Cue Exposure; Behavioral: Progressive Muscle Relaxation; Drug: Placebo

INTERVENTIONS:
Drug: D-cycloserine
  Arms: D-cycloserine
Drug: Nicotine Replacement Therapy (patch)
Behavioral: Smoking Cue Exposure
Behavioral: Progressive Muscle Relaxation
Drug: Placebo — The investigators will administer Gelatin Capsule instead of D-Cycloserine in a double blind fashion to some of study subjects.
  Arms: Gelatin Capsule

SUMMARY:
The investigators previously developed a cigarette cue extinction treatment (CET) procedure in non-treatment seeking volunteer smokers in our nicotine laboratory. The goal of Cue Extinction Treatment is to un-pair a behavioral or autonomic response from the stimulus that triggers it. This is accomplished through repeated exposure to that trigger, while removing the patient's ability to act out the conditioned response. In the present study, the trigger is a lit cigarette, and the response the investigators seek to un-pair is cigarette craving. In the procedure the investigators have previously developed and intend to use again, the participant is shown a pack of his brand of choice cigarettes. The researcher removes a cigarette from the pack, lights it, and asks the participant to hold the cigarette without smoking it for 90 seconds. This procedure is repeated seven times over the course of a six-hour lab session. The investigators hope to boost the clinical response to smoking cue exposure therapy in quitters on NRT (nicotine replacement therapy) pretreatment by pharmacological augmentation with the partial NMDA receptor agonist D-cycloserine (DCS). Behavioral extinction training is a form of learning that may be modulated by NMDA receptor mediated glutamate transmission. The study's main hypothesis is that the partial NMDA receptor agonist D-cycloserine (DCS) facilitates cue exposure training and may prevent relapse to smoking. The aim of the proposed study is to assess whether DCS-facilitation of cue-exposure therapy improves abstinence among smokers on the nicotine patch seeking treatment. Development of an effective treatment strategy to enhance the effectiveness of NRTs would have a direct and significant positive impact on public health.

ELIGIBILITY:
Inclusion Criteria:

1. Seeking treatment for nicotine dependence
2. Medically healthy on the basis of physical examination and medical history, vital signs, EKG, and laboratory tests, with a negative pregnancy test for females.
3. A DSM-IV diagnosis of nicotine dependence with physiological dependence. Has smoked at least 15 cigarettes daily for at least two years.
4. Able to perform study procedures.
5. Males or females between the ages of 21-55 yrs.
6. Female Participants agree to use an effective method of birth control

Exclusion Criteria:

1. A DSM-IV diagnosis of lifetime history of abuse or dependence on alcohol or drugs other than nicotine
2. Current Axis I diagnosis or current treatment with psychotropic medications (within last three months).
3. Lifetime history of schizophrenia or other psychotic disorders, bipolar disorder, or anxiety disorders.
4. Participants on parole or probation
5. History of significant recent violent behavior, e.g., one or more incidents of violent behavior in the past year resulting in physical damage.
6. Unstable medical condition, Blood pressure > 140/90, Pregnancy.
7. History of allergic reaction to nicotine patch.
8. History of hypersensitivity to cycloserine.
9. Any history of seizures
10. History of renal disease.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of Cigarettes Smoked | 3 months
  Smoking Diary kept of daily cigarette smoking.

CONTACTS AND LOCATIONS:
Overall Officials: S. Rob Vorel, MD, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States